CLINICAL TRIAL: NCT03658148
Title: Association Between Hematological Ratios and Acute Kidney Injury After Cardiovascular Surgery in Neonates: a Retrospective Observational Study
Brief Title: Hematologic Ratios in Postoperative Acute Kidney Injury
Status: Withdrawn | Type: Observational
Why Stopped: No charts were reviewed. This study never started.
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Responsible Party: Sponsor
Other Study IDs: CIN001-AKI Hematologic Ratios
Record Dates: First submitted 2018-08-06; First posted 2018-09-05 (Actual); Last update posted 2024-11-06 (Actual); Status verified 2021-06

CONDITIONS: Acute Kidney Injury
Keywords: Acute Kidney Injury; Cardiac Surgery; Cardiopulmonary Bypass; Congenital Heart Disease; Biomarkers
MeSH Terms: conditions — Acute Kidney Injury; Heart Defects, Congenital | interventions — Cardiac Surgical Procedures; Cardiopulmonary Bypass

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Study Group: Neonates (≤31 days) who underwent cardiac surgery with cardiopulmonary bypass for congenital heart disease (CHD) between 2008-2017.
  Interventions: Procedure: Cardiac Surgery with Cardiopulmonary Bypass

INTERVENTIONS:
Procedure: Cardiac Surgery with Cardiopulmonary Bypass — Cardiac Surgery with Cardiopulmonary Bypass

SUMMARY:
Acute kidney injury (AKI) is a common complication after surgery for congenital heart disease and is associated with significant morbidity and mortality. To-date, no biomarker has been universally implemented for predicting AKI in neonates after cardiac surgery. In this study, the use of hematological ratios will be evaluated for predicting AKI and postoperative outcomes in this patient cohort.

DETAILED DESCRIPTION:
In adults, hematological ratios which can be calculated from a routinely ordered complete blood count with differential, such as the neutrophil/lymphocyte ratio, have been demonstrated to be correlated with acute kidney injury (AKI) and other clinical outcomes after cardiovascular surgery. In this retrospective observational study, the association between hematological ratios (neutrophil/lymphocyte ratio, platelet/lymphocyte ratio, neutrophil/lymphocyte*platelet ratio, monocyte/lymphocyte ratio, and plateletcrit) and postoperative AKI, morbidity (length of ICU stay, hospital stay, mechanical ventilation, vasoactive infusion-free days, etc.) and mortality will be evaluated in neonates who underwent cardiac surgery with cardiopulmonary bypass.

ELIGIBILITY:
Inclusion Criteria:

* Neonates (≤31 days) who underwent cardiac surgery with cardiopulmonary bypass for congenital heart disease.

Exclusion Criteria:

* Patients with missing relevant preoperative or postoperative data points
* Patients with previous palliation or reoperation,
* Thymus hypo/aplasia (DiGeorge Syndrome, Ataxia-telangiectasia, or Nezelof syndrome),
* Primary immunodeficiency,
* Episode of cardiac arrest within 1 week before surgery,
* Signs or history of preoperative renal impairment or AKI (KDIGO Stage ≥1 observed on preoperative labs),
* Hypothyroidism,
* Patients with a history of infection within a week prior to surgery or antibiotics administered within the first 3 days after surgery (except for postoperative antibiotics).

Ages: 0 Days to 31 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Neonates (≤31 days) who underwent cardiac surgery with cardiopulmonary bypass for congenital heart disease between 2008-2017.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2018-07-01 (Actual); Primary Completion 2020-11-01 (Actual); Study Completion 2021-06-01 (Actual)

PRIMARY OUTCOMES:
Acute Kidney Injury (AKI) | up to 72 hours postoperative
  Occurrence of AKI as defined by the Kidney Disease Improving Global Outcomes (KDIGO) diagnostic classification (using serum creatinine)

SECONDARY OUTCOMES:
Operative Mortality | up to 30 days postoperative
  Mortality within 30 days after surgery (rate)
1-year mortality | up to 1 year postoperative
  Mortality within 1 year after surgery (rate)
Length of hospital stay | up to 1 year postoperative
  Total length of hospital stay (days)
Length of Cardiac Intensive Care Unit (CICU) Stay | up to 1 year postoperative
  Total length of stay in the CICU (days)
Length of mechanical ventilation | up to 1 year postoperative
  Total length of postoperative mechanical ventilator support (days)
Vasoactive infusion-free days | up to 28 days postoperative
  (days)
Postoperative infection | up to 3 days postoperative
  Occurrence of infection defined as: antibiotic use (other than perioperative) within 3 days postop, positive blood culture within 3 days postop, positive viral panel within 3 days postop
Low Cardiac Output Syndrome | up to 2 days postoperative
  Occurrence of Low Cardiac Output Syndrome defined as any of the following at any time during the first 48 hours postoperative:
  1. Lactate >6mmol/l and mixed venous saturation (ScvO2) <60% (or SaO2-ScvO2 difference greater than 35% in a single ventricle),
  2. Vasoactive inotropic score (VIS)3 ≥ 10,
  3. Extracorporeal Membrane Oxygenation (ECMO

CONTACTS AND LOCATIONS:
Locations (1):
- Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio, United States

IPD SHARING:
Plan to Share IPD: No